CLINICAL TRIAL: NCT06660888
Title: Study of Chronic Fatigue, Depression, and Anxiety Among Hypothyroid Patients Attending Assuit University Hospitals
Status: Enrolling by invitation | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Hamdy Rashed, Resident Doctor at Family Medicine Department, Assiut University
Other Study IDs: Fatigue in Hypothyroidism
Record Dates: First submitted 2024-10-10; First posted 2024-10-28 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Hypothyroidism Primary
Keywords: Fatigue; Depression; Anxiety
MeSH Terms: conditions — Hypothyroidism; Fatigue; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: • Fatigue Severity Scale (FFS). • Hamilton Rating Scale for Depression (HRSD-17). • Hamilton Anxiety Rating Scale (HAM-A). — 1. Fatigue Severity Scale The FSS is one of the most commonly used fatigue questionnaires in chronic diseases. It measures how fatigue affects motivation, exercise, physical functioning, carrying out duties, work, family, or social life.
  2. Hamilton Depression Rating Scale The 17-item Hamilton Depression Rating Scale (HRSD-17) is the most popular depression measure in antidepressant clinical trials.
  3. Hamilton Anxiety Rating Scale The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms.

SUMMARY:
* Assessment of the prevalence of chronic fatigue, depression, and anxiety among patients with hypothyroidism in Assuit University Hospital.
* Assess the severity of chronic fatigue, depression, and anxiety according to the duration and control of treatment in patients with hypothyroidism.

DETAILED DESCRIPTION:
Hypothyroidism is a prevalent endocrine illness with a global impact, necessitating treatment in extreme instances. Inadequate management of hypothyroidism has been associated with adverse health outcomes, including neurological and musculoskeletal issues,this condition impacting approximately 1-6% of the general population.

Thyroid hormone is essential for the normal development of many human tissues and regulates the metabolism of virtually all cells and organs of the human body throughout life. Overt hypothyroidism is defined by thyroid-stimulating hormone (TSH) levels above the upper limit of the reference range, while levels of free thyroxine (fT4) are below the lower limit of the reference range. The reference range is typically statistically defined by the 2.5th and 97.5th percentiles of the measured circulating thyroid hormone values in populations defined as healthy.

It has been reported that up to one-third of patients presenting with fatigue have thyroid disease, predominantly in women,and fatigue was the most common noted symptom among patients with hypothyroidism.Also patients with thyroid disorders are more prone to developing depressive symptoms.

There are few previous studies that addressed this topic in the Egyptian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary hypothyroidism.
* Age from 18 to 60 years.

Exclusion Criteria:

* Patients who were previously diagnosed with any psychiatric diseases.
* Serious and chronic diseases (e.g. anemia, liver, heart or kidney problems).
* consumption of medications that may interfere with thyroid function (e.g., chemotherapy), patients who had a history of any type of cancer, due to the confounding effects of cancer on fatigue as the outcome of interest.
* Women who were pregnant or had given birth in the last 6 months to exclude postpartum thyroiditis and depression.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with primary hypothyroidism with age from 18 to 60 years.
Sampling Method: Non-Probability Sample
Enrollment: 406 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of chronic fatigue in patients with hypothyroidism at Assuit University Hospitals. | Baseline
  Prevelance of fatigue will be assessd by fatigue severity scale, this scale consists of nine items, each item consists of statements that are scored on a seven-point Likert type scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The minimum score is 9 and the maximum score possible is 63. Higher the score = greater fatigue severity.
  The scores are averaged across the nine statements, and a score ≥36 indicates a clinically significant trait level of fatigue.
Prevalence of depression in patients with hypothyroidism at Assuit University Hospitals. | Baseline
  Prevalence of depression will be assessed by Hamilton Rating Scale for Depression ,it consists of 17 items, each of them is rated on a 0-4 scale, except for items 10 (sleep disorders) and 14 (somatic symptoms), which are rated on a 0-2 scale. The scores are interpreted as follows :
  HAM-D score 7-17: mild depression; HAM-D score 18-24: moderate depression; and HAM-D score 25 or higher: severe depression
Prevalence of anxiety in patients with hypothyroidism at Assuit University Hospitals. | Baseline
  Prevalence of anxiety will be assessed by Hamilton Rating Scale of Anxiety, The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
  Each item is scored on a scale of 0 (not present) to 4 (very severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

SECONDARY OUTCOMES:
Compare the severity of chronic fatigue according to the duration and control of treatment in patients with hypothyroidism. | Baseline
  By using the Fatigue Severity Scale with the minimum score is 9 and the maximum score possible is 63. The higher the score the greater fatigue severity.
  We will compare the severity of fatigue to the duration of levothyroxine treatment and if there is improvement of fatigue severity in hypothyroidism patients with good control of treatment or not.
Compare the severity of depression according to the duration and control of treatment in patients with hypothyroidism. | Baseline
  By using the Hamilton Depression Rating Scale with the following scores; HAM-D score 7-17: mild depression; HAM-D score 18-24: moderate depression; and HAM-D score 25 or higher: severe depression. We will compare the relationship between the severity of depression and the duration and control of levothyroxine treatment in hypothyroid patients.
  We will compare if there is improvement of the severity of depression with good control of treatment or not.
Compare the severity of anxiety according to the duration and control of treatment in patients with hypothyroidism. | Baseline
  By using the Hamilton Anxiety Rating Scale with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. We will compare the relationship between the severity of anxiety and the duration of levothyroxine treatment in hypothyroid patients and if there is improvement of anxiety with good control of treatment or not.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Elkhateeb, Prof., Study Director — Assiut University; Romany H Gabra, A prof., Study Director — Assiut University; Dalia G Mohammed, Prof., Study Director — Assiut University
Locations (1):
- Assuit university hospitals, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Udovcic M, Pena RH, Patham B, Tabatabai L, Kansara A. Hypothyroidism and the Heart. Methodist Debakey Cardiovasc J. 2017 Apr-Jun;13(2):55-59. doi: 10.14797/mdcj-13-2-55. PMID 28740582
- [Background] Sethi B, Barua S, Raghavendra MS, Gotur J, Khandelwal D, Vyas U. The Thyroid Registry: Clinical and Hormonal Characteristics of Adult Indian Patients with Hypothyroidism. Indian J Endocrinol Metab. 2017 Mar-Apr;21(2):302-307. doi: 10.4103/ijem.IJEM_387_16. PMID 28459030
- [Background] Evans KM, Flanagan DE, Wilkin TJ. Chronic fatigue: is it endocrinology? Clin Med (Lond). 2009 Feb;9(1):34-8. doi: 10.7861/clinmedicine.9-1-34. PMID 19271598
- [Background] Ruiz-Pacheco MG, Hernandez I, Hernandez-Estrella G, Basurto L, Vargas-Ortega G, Gonzalez-Virla B, Molina-Ayala M, Hernandez-Martinez AF, Luengas-Mondragon R, Hernandez-Allende AA, Mendoza-Zubieta V, Balcazar-Hernandez L. Severity of Fatigue and Its Relationship with TSH before and after Levothyroxine Replacement Therapy in Patients with Primary Hypothyroidism. Biomedicines. 2023 Mar 7;11(3):811. doi: 10.3390/biomedicines11030811. PMID 36979787
- [Background] Chaker L, Razvi S, Bensenor IM, Azizi F, Pearce EN, Peeters RP. Publisher Correction: Hypothyroidism. Nat Rev Dis Primers. 2022 Jun 10;8(1):39. doi: 10.1038/s41572-022-00373-7. No abstract available. PMID 35688906
- [Background] Nassar M, Hassan A, Ramadan S, Desouki MT, Hassan MA, Chaudhuri A. Evaluating the effectiveness of combined T4 and T3 therapy or desiccated thyroid versus T4 monotherapy in hypothyroidism: a systematic review and meta-analysis. BMC Endocr Disord. 2024 Jun 14;24(1):90. doi: 10.1186/s12902-024-01612-6. PMID 38877429
- [Background] Ali ZH, Abdulridha MK, Alzajaji QB. Screening factors affecting proper levothyroxine therapy among patients with primary hypothyroidism: a cross-sectional study. J Med Life. 2024 Feb;17(2):177-187. doi: 10.25122/jml-2023-0387. PMID 38813351
- [Background] Hage MP, Azar ST. The Link between Thyroid Function and Depression. J Thyroid Res. 2012;2012:590648. doi: 10.1155/2012/590648. Epub 2011 Dec 14. PMID 22220285